CLINICAL TRIAL: NCT02801162
Title: Evaluation of Accuracy and Precision of the Proxima 3® (Sphere Medical) Arterial Blood Gas Analysis System in Comparison With the Reference Standard Hospital ABG in a Rapidly Changing Clinical Context
Brief Title: Evaluation of Accuracy and Precision of a New Arterial Blood Gas Analysis System Blood in Comparison With the Reference Standard
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: To much effort needed, high costs for an academic study
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PROXIMA
Record Dates: First submitted 2016-05-31; First posted 2016-06-15 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2018-10

CONDITIONS: Hypoxia; Hypercapnia; Anaemia
Keywords: arterial blood gas
MeSH Terms: conditions — Hypoxia; Hypercapnia; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional ABG analyser (Active Comparator)
  Interventions: Device: conventional ABG analyser; Device: Proxima 3®
- Proxima 3® arterial blood gas (Experimental)
  Interventions: Device: conventional ABG analyser; Device: Proxima 3®

INTERVENTIONS:
Device: conventional ABG analyser — pO2 mmHg, pH, pCO2 mmHg, Base excess, Hct %
Device: Proxima 3® — pO2 mmHg, pH, pCO2 mmHg, Base excess, Hct %

SUMMARY:
Evaluate the precision and accuracy of the Proxima 3® System by obtaining quantitative clinical data at various time points. Compare the methods associated with obtaining blood gas results using the Proxima 3® System device versus a conventional ABG analyse. The aim of the investigator is to evaluate the precision and accuracy of the Proxima 3® ABG system parameters (pH, pCO2 pO2, hematocrit and potassium) in clinical practices with rapid changing context.

DETAILED DESCRIPTION:
In this study the investigator will test the applicability of the Proxima 3® ABG system in a heterogeneous patient population consisting of patients scheduled for hybrid atrial fibrillation surgery, patients scheduled for heart valve surgery, complex cardiac surgery with deep cooling, spine surgery or patients with expected major blood loss. The investigator will compare the ABG values obtained with the traditional ABG measurement system of the hospital.

The availability of a disposable patient-dedicated blood gas analyser allows rapid, frequent measurement of blood gases in theatre without the loss of theatre staff. As well as facilitating measurement in the unstable patient, this approach opens up the possibility for more frequent measurement to identify patient deterioration before a crisis occurs.

The conventional laboratory ABG method uses sensor technology for pH, pCO2, pO2, sodium, potassium, calcium, glucose and lactate levels. It measures hemoglobin concentration via spectrophotometry methodology at a set wavelength of 467-672 nm. The blood gas laboratory uses ABL90 Flex (Radiometer®). The optical system is based on a 138-wavelength spectrophotometer with a measuring range of 467-672 nm. The spectrophotometer is connected via an optical fiber to a combined hemolyzer and measuring chamber.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years old
* Patients who have (or will have) an arterial line, which was (will be) inserted for clinical - need, will be considered for inclusion in this study
* Patients who give informed consent (or their personal/nominated consultee) to participate in the study
* Patients who are likely to have an arterial line for at least 6 hours.

Exclusion Criteria:

* Patients contraindicated for an arterial line
* Refusal of consent by a patient
* Not for use with patients with uncorrected hyperphosphataemia, hypocalcaemia or hypercalcaemia.
* The patient is considered to be unsuitable for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of accuracy and precision of the Proxima 3® for ABG | From intubation until extubation, max 1 day
  Evaluate the precision and accuracy of the Proxima 3® System by obtaining quantitative clinical data at various time points

SECONDARY OUTCOMES:
Time to obtain an arterial blood gas | From intubation until extubation, max 1 day
  Time for obtaining arterial blood gas: prelevation time to result time

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Umbrain, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel; Jan Poelaert, MD, PhD, Study Director — Universitair Ziekenhuis Brussel; Manuella Martin, Apr. Biol., Study Chair — Universitair Ziekenhuis Brussel; Christine Sneyers, Nurse, Principal Investigator — Universitair Ziekenhuis Brussel; Gabriel Kotolácsi, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Pierre Matagne, Nurse, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes